CLINICAL TRIAL: NCT01992341
Title: An Open-Label, Pharmacokinetic Drug-Drug Interaction (DDI) Study of AMG 386 in Combination With Paclitaxel in Adult Subjects With Advanced Solid Tumors
Brief Title: AMG 386 Drug-Drug Interaction Study With Paclitaxel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20101151
Record Dates: First submitted 2012-06-14; First posted 2013-11-25 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Advanced Solid Tumors
Keywords: sarcomas; carcinomas
MeSH Terms: conditions — Sarcoma; Carcinoma | interventions — trebananib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AMG 386 15mg/kg and paclitaxel 80mg/m2 (Experimental)
  Interventions: Drug: AMG 386; Drug: Paclitaxel

INTERVENTIONS:
Drug: AMG 386 — Weekly 15 mg/kg of AMG 386 in combination with three weeks on/ one week off 80mg/m2 of paclitaxel. Continued therapy with AMG 386 with or without paclitaxel until progression, unacceptable toxicity develops, or study withdrawal.
  Other Names: Taxol
Drug: Paclitaxel — Three weeks on/ one week off 80mg/m2 of paclitaxel in combination with weekly 15 mg/kg of AMG 386 . Continued therapy with AMG 386 until progression, unacceptable toxicity develops, or study withdrawal. A cycle consists of 3 weeks on / 1 week off of paclitaxel.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of paclitaxel when given alone and in combination with AMG 386 to determine whether AMG 386 alters the pharmacokinetics of paclitaxel

DETAILED DESCRIPTION:
Eligible subjects enrolled in the study will begin receiving paclitaxel on a three weeks on / one week off schedule at study day 1 and weekly AMG 386 beginning at study day 8. The pharmacokinetic portion of the study occurs during the first two study cycles with intensive PK collections on study weeks 1, 6 and 8. Once the pharmacokinetic assessment period is completed, continued combination therapy with AMG 386 and paclitaxel or single-agent AMG 386 will be administered at the investigator's discretion until progression, unacceptable toxicity develops, or study withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years of age
* Have a pathologically documented, and definitely diagnosed, advanced solid tumor that is refractory to standard treatment, or for which no curative therapy is available
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Normal or clinically acceptable ECG (12 lead reporting PR, QRS, QTc)

Exclusion Criteria:

* Subjects with gastric cancer or any malignancy with purely squamous cell histology
* Known history of primary central nervous system (CNS) tumors or CNS metastases
* Myocardial infarction within 1 year before study day 1, unstable or uncontrolled disease/condition related to or affecting cardiac function
* History of stroke, arterial or venous thrombosis, or pulmonary embolism within 1 year before study day 1
* A baseline ECG QTc interval > 450 msec
* Active grade 2 or greater peripheral vascular disease
* History of pulmonary hemorrhage or gross hemoptysis within 6 months before study day 1
* Non-healing wound, ulcer (including gastrointestinal) or fracture
* Known positive test for human immunodeficiency virus infection, or active hepatitis B or hepatitis C infection
* Major surgery within 1 month before study day 1
* Concurrent antitumor treatment within 4 weeks (6 weeks for nitrosoureas or mitomycin) before study day 1
* Unable to tolerate IV administration or repeated blood withdrawal
* Hypersensitivity to paclitaxel or drugs using the vehicle cremophor
* Known sensitivity to mammalian-derived products, bacterially-produced proteins, or any of the products to be administered during dosing
* Chronic neuropathy grade ≥ 1
* Concurrent or prior treatment with 2C8 and 3A4 substrates
* Enrolled in or has not yet completed at least 30 days (prior to study day 1) since ending other investigational device or drug, or currently receiving other investigational treatment.
* Men and woman of reproductive potential, unwilling to practice a highly effective method of birth control for the duration of the study and an additional 6 months after the last dose of AMG 386
* Women who are lactating/breastfeeding
* Women with a positive pregnancy test
* Women planning to become pregnant during the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Paclitaxel PK parameters | 9 weeks
  Paclitaxel PK parameters with and without the co-administration of AMG 386.

SECONDARY OUTCOMES:
AMG 386 PK parameters | 9 weeks
  AMG 386 PK steady state PK parameters with and without paclitaxel co-administration
Safety | Average of 6 months
  Subject incidence of treatment-emergent adverse events: Assessments include physical examinations, vitals, clinical laboratories, and electrocardiograms (ECG) • Results of safety laboratory tests, vital sign measurements, and ECG measurments
Safety | Average of 6 months
  Incidence of anti-AMG 386 antibody formation

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com